CLINICAL TRIAL: NCT03342274
Title: Adapting the Diabetes Prevention Program for a Developing World Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of the Western Cape (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15080328
Record Dates: First submitted 2017-11-10; First posted 2017-11-14 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: After the end of year 1 outcomes the control arm crosses over and a year 2 follow-up is conducted on both arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Program Intervention (Experimental): Participants receive usual care and group weight loss sessions adapted from the Diabetes Prevention Program delivered by Community Health Workers.
  Interventions: Behavioral: Lifestyle Program; Other: Usual Care
- Wait list (Other): Participants receive usual care and after 1 year receive the Lifestyle Program intervention
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Lifestyle Program — Participants will receive group weight loss sessions addressing healthy eating, exercise, and weight loss principles adapted from the Diabetes Prevention Program delivered by Community Health Workers.
  Arms: Lifestyle Program Intervention
Other: Usual Care — Usual care consists of chronic disease management through medication delivery and monitoring of weight, blood pressure, and blood glucose by Community Health Workers.

SUMMARY:
This study will examine whether an adapted version of ]he Diabetes Prevention Program (DPP) can be effective when delivered by community health workers (CHWs) in a poor urban community in South Africa. We will randomize existing groups that are part of an non-governmental organization's (NGO) chronic disease management program (anticipated cluster N = 54; anticipated individual N=540), to receive either the program or usual care (wait-list). The primary outcome analysis will compare percentage of baseline weight loss at Y1 between the program and usual care; however, after Y1 usual care participants will also receive the program and both groups will be followed for another year.

ELIGIBILITY:
Inclusion Criteria:

* member of participating partner NGO "health club" (members are medically stabilized individuals with diabetes mellitus or hypertension referred for disease and lifestyle management)
* BMI greater than or equal to 25 kg per meter squared

Exclusion Criteria:

* unsafe level of blood pressure (greater than or equal to 160 (systolic) and greater than equal to 100 mm (diastolic)) at screening
* elevated blood sugar (A1C greater than 11) at screening
* being pregnant, breast-feeding or planning pregnancy within 2 years
* chronic use of oral steroid medication
* intellectual disabilities that would prevent ability to understand the program
* not intending to stay in the health club over the next 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Weight loss | 1 year
  percentage weight loss (weight measured in kilograms)

SECONDARY OUTCOMES:
Blood pressure | 1 year
  systolic blood pressure (mmHG), diastolic blood pressure (mmHG)
HbA1c | 1 year
  percent
LDL cholesterol | 1 year
  mg/dl
Triglycerides | 1 year
  mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Western Cape, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Materia FT, Smyth JM, Puoane T, Tsolekile L, Goggin K, Kodish SR, Fox AT, Resnicow K, Werntz S, Catley D. Implementing text-messaging to support and enhance delivery of health behavior change interventions in low- to middle-income countries: case study of the Lifestyle Africa intervention. BMC Public Health. 2023 Aug 10;23(1):1526. doi: 10.1186/s12889-023-16388-y. PMID 37563595
- [Derived] Whittington MD, Goggin K, Tsolekile L, Puoane T, Fox AT, Resnicow K, Fleming KK, Smyth JM, Materia FT, Hurley EA, Vitolins MZ, Lambert EV, Levitt NS, Catley D. Cost-effectiveness of Lifestyle Africa: an adaptation of the diabetes prevention programme for delivery by community health workers in urban South Africa. Glob Health Action. 2023 Dec 31;16(1):2212952. doi: 10.1080/16549716.2023.2212952. PMID 37220094
- [Derived] Catley D, Puoane T, Tsolekile L, Resnicow K, Fleming KK, Hurley EA, Smyth JM, Materia FT, Lambert EV, Vitolins MZ, Levitt NS, Goggin K. Evaluation of an adapted version of the Diabetes Prevention Program for low- and middle-income countries: A cluster randomized trial to evaluate "Lifestyle Africa" in South Africa. PLoS Med. 2022 Apr 15;19(4):e1003964. doi: 10.1371/journal.pmed.1003964. eCollection 2022 Apr. PMID 35427357
- [Derived] Catley D, Puoane T, Tsolekile L, Resnicow K, Fleming K, Hurley EA, Smyth JM, Vitolins MZ, Lambert EV, Levitt N, Goggin K. Adapting the Diabetes Prevention Program for low and middle-income countries: protocol for a cluster randomised trial to evaluate 'Lifestyle Africa'. BMJ Open. 2019 Nov 11;9(11):e031400. doi: 10.1136/bmjopen-2019-031400. PMID 31719084